CLINICAL TRIAL: NCT03637335
Title: Phase-3 Study, Randomized, Controlled, Multi-center, Double Blind, Comparing Palliative Radiotherapy With or Without Carboplatin
Brief Title: Comparing Palliative Radiotherapy With or Without Carboplatin
Acronym: METAXIOM
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The study was stopped due to insufficient recruitment.
Sponsor: Institut Cancerologie de l'Ouest (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ICO-A-2014-11
Record Dates: First submitted 2018-08-06; First posted 2018-08-20 (Actual); Last update posted 2018-08-20 (Actual); Status verified 2018-07

CONDITIONS: Lung Cancer; Head and Neck Cancer; Metastatic Cancer
Keywords: irradiation; placebo; carboplatin
MeSH Terms: conditions — Lung Neoplasms; Head and Neck Neoplasms; Neoplasm Metastasis | interventions — Radiation; Carboplatin

STUDY DESIGN:
Intervention Model Description: Phase-3 study, randomized, controlled, multi-center, double blind
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- irradiation + carboplatin (Experimental): Radiotherapy in 30 Gy en 10 fractions de 3 Gy. The overall duration to irradiation is 2 weeks Carboplatin. :10 injections 1h prior irradiation
  Interventions: Combination Product: irradiation + carboplatin
- irradiation + placebo (Placebo Comparator): Radiotherapy in 30 Gy en 10 fractions de 3 Gy. The overall duration to irradiation is 2 weeks Placebo :10 injections 1h prior irradiation
  Interventions: Combination Product: irradiation + placebo

INTERVENTIONS:
Combination Product: irradiation + carboplatin — 30 Gy en 10 fractions de 3 Gy + 10 injections of carboplatin
  Arms: irradiation + carboplatin
Combination Product: irradiation + placebo — 30 Gy en 10 fractions de 3 Gy + 10 injections of placebo
  Arms: irradiation + placebo

SUMMARY:
The study population has locally advanced or metastatic bronchial or head and neck cancer.

This study assesses the value of concomitant chemo/radiotherapy with carboplatin daily during metastatic radiotherapy versus radiotherapy alone.

The realization of a systemic treatment during the radiotherapy could make it possible to obtain a benefit on the control of the evolution of the metastases and thus of the pains generated, as well as on the quality of life of the patients. In addition, a benefit in overall survival is possible.

DETAILED DESCRIPTION:
The study population has locally advanced or metastatic bronchial or head and neck cancer.

Patients receive 10 injections of carboplatin (validated chemo-sensitizing molecule) or placebo (glucose) before 10 radiation sessions.

The overall duration is 14 days.

ELIGIBILITY:
Inclusion Criteria:

* Patients with locally advanced or metastatic bronchial or head and neck cancer
* Patient require palliative radiotherapy
* Age ≥ 18 years
* PS ≤ 2
* Obtaining the signed written consent of the patient
* Patient affiliated to a social security scheme

Exclusion Criteria:

* Other chemotherapy or targeted therapy
* Prior radiation
* Patients with thrombopenia < 100 000
* Patients with neutropenia < 2000
* Patients with renal clearance < 20 mL/min
* Known hypersensitivity to platinum salt
* Treatment with phenytoin or fosphenytoin
* In previous three months, a vaccination against yellow fever, live vaccin or live attenuated vaccine
* Unchecked diabetes
* hemorrhagic tumor
* Refusal of participation or inability to issue informed consent
* Person deprived of liberty or adult under guardianship
* Minor patients, pregnant or lactating women
* Participation in other interventional study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2015-08-17 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2018-05-28 (Actual)

PRIMARY OUTCOMES:
Local progression-free survival of chemo radiotherapy compared with placebo-associated radiotherapy | 36 months
  = delay between the start date of treatment and the date of the first event related to the treated location

SECONDARY OUTCOMES:
Impact in quality of life | 25 months
  Evaluate with questionnaire QLQ-C30 at inclusion, at the end of treatment and during the following
Variation in intensity of pain | 25 months
  Analogical visual scale (EVA)
evolution of dose of pain medication | 25 months
  variation of dosage of pain medication between inclusion and the end of radiotherapy (mg, number of caps, ...)
toxicity due to radiotherapy | 25 months
  Toxicity 4 weeks after radiotherapy with NCI-CTC-AE v4
overall survey | 36 months
  Time between inclusion and death
To evaluate free progression survival | 36 months
  Time between inclusion and first progression

CONTACTS AND LOCATIONS:
Overall Officials: FABRICE DENIS, MD, Principal Investigator — Centre Jean Bernard
Locations (2):
- France (2):
  - Fabrice Denis, Le Mans
  - Institut de Cancérologie de l'Ouest, Nantes

IPD SHARING:
Plan to Share IPD: No